CLINICAL TRIAL: NCT00262470
Title: Treatment of Orthostatic Intolerance
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Satish R. Raj (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Satish R. Raj, Assistant Professor of Medicine & Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 008397; UL1TR000445 (NIH)
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Tachycardia; Chronic Orthostatic Intolerance
Keywords: tachycardia; sinus tachycardia; postural tachycardia syndrome (POTS)
MeSH Terms: conditions — Tachycardia; Tachycardia, Sinus; Postural Orthostatic Tachycardia Syndrome | interventions — Acetazolamide; Atomoxetine Hydrochloride; Clonidine; entacapone; Propranolol; Indomethacin; Mecamylamine; Isosorbide Dinitrate; Melatonin; Midodrine; Modafinil; Octreotide; Sertraline; Sodium Chloride; Saline Solution; Drinking Water; Memantine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (20):
- 1 (Experimental): Acetazolamide
  Interventions: Drug: Acetazolamide
- 2 (Experimental): Atomoxetine
  Interventions: Drug: Atomoxetine; Drug: Atomoxetine & Propranolol
- 3 (Experimental): NO Drug
  Interventions: Other: NO Drug
- 4 (Experimental): Clonidine
  Interventions: Drug: Clonidine
- 5 (Experimental): Entacapone
  Interventions: Drug: Entacapone; Drug: Entacapone & Propranolol
- 6 (Experimental): Indomethacin
  Interventions: Drug: Indomethacin
- 7 (Experimental): Isosorbide Dinitrate
  Interventions: Drug: Isosorbide Dinitrate
- 8 (Experimental): Mecamylamine
  Interventions: Drug: Mecamylamine
- 9 (Experimental): Memantine
  Interventions: Drug: memantine
- 10 (Experimental): Melatonin
  Interventions: Dietary Supplement: Melatonin
- 11 (Experimental): Midodrine
  Interventions: Drug: Midodrine
- 12 (Experimental): Modafinil
  Interventions: Drug: Modafinil; Drug: Modafinil & Propranolol
- 13 (Experimental): Octreotide
  Interventions: Drug: Octreotide
- 14 (Placebo Comparator): Placebo (lactose tablet)
  Interventions: Radiation: Placebo
- 15 (Experimental): Propranolol
  Interventions: Drug: Entacapone & Propranolol; Drug: Atomoxetine & Propranolol; Drug: Propranolol; Drug: Modafinil & Propranolol
- 16 (Experimental): Sertraline
  Interventions: Drug: Sertraline
- 17 (Experimental): Normal Saline (0.9%) 1 liter
  Interventions: Procedure: IV Saline
- 18 (Experimental): Drinking Water
  Interventions: Other: Drinking Water
- 19 (Experimental): Dead Space Breathing Device
  Interventions: Device: Breathing Device
- Abdominal Binder (Experimental): Abdominal binder with inflatable pressure over abdomen
  Interventions: Device: Abdominal binder

INTERVENTIONS:
Drug: Acetazolamide — 250 mg PO x 1
  Other Names: Diamox
  Arms: 1
Drug: Atomoxetine — 10-40 mg PO x 1 dose
  Other Names: Strattera
  Arms: 2
Other: NO Drug — No intervention - just monitoring
  Arms: 3
Drug: Clonidine — Clonidine 0.05-0.3 mg PO x 1 dose
  Other Names: Catapres
  Arms: 4
Drug: Entacapone — Entacapone 200-400 mg PO x 1 dose
  Other Names: Comtan
  Arms: 5
Drug: Entacapone & Propranolol — Entacapone 200-400 mg PO x 1 dose AND propranolol 20 mg PO x 1 dose
  Other Names: Comtan; Inderal
  Arms: 15; 5
Drug: Atomoxetine & Propranolol — Atomoxetine 10-40 mg PO x 1 dose AND propranolol 20 mg PO x 1 dose
  Other Names: Strattera; Inderal
  Arms: 15; 2
Drug: Indomethacin — Indomethacin 25-50 mg PO x 1 dose
  Other Names: Indocin
  Arms: 6
Drug: Mecamylamine — mecamylamine 1.25-5 mg PO x 1 dose
  Other Names: inversine
  Arms: 8
Drug: Isosorbide Dinitrate — Isosorbide dinitrate 5-20 mg PO x 1 dose
  Other Names: Isordil
  Arms: 7
Dietary Supplement: Melatonin — melatonin 3 mg PO x 1 dose
  Arms: 10
Drug: Midodrine — midodrine 2.5-10 mg PO x 1 dose
  Other Names: pro-amatine
  Arms: 11
Drug: Modafinil — modafinil 100-200 mg PO x 1 dose
  Other Names: provigil
  Arms: 12
Drug: Octreotide — octreotide 12.5-50 mcg Subcutaneous x 1 dose
  Other Names: sandostatin
  Arms: 13
Radiation: Placebo — lactose tablet x 1 pill
  Arms: 14
Drug: Propranolol — Propranolol 10-80 mg PO x 1-2 dose
  Other Names: Inderal
  Arms: 15
Drug: Modafinil & Propranolol — Modafinil 100-200 mg PO x 1 dose AND Propranolol 20 mg PO x 1 dose
  Other Names: Provigil; Inderal
  Arms: 12; 15
Drug: Sertraline — sertraline 25-50 mg PO x 1 dose
  Other Names: Zoloft
  Arms: 16
Procedure: IV Saline — 1 liter IV over 2 hours
  Other Names: NaCl solution (0.9%)
  Arms: 17
Other: Drinking Water — 16 fluid ounces
  Arms: 18
Device: Breathing Device — Breathing through a dead space tube
  Arms: 19
Drug: memantine — memantine 5-20 mg PO x 1 dose
  Other Names: Namenda
  Arms: 9
Device: Abdominal binder — Using large blood pressure cuffs linked together, they are wrapped around the subjects abdomen and inflated to generate increased pressure to below tolerably threshold.
  Arms: Abdominal Binder

SUMMARY:
This trial is designed to study the effects of various mechanistically unique medications in controlling excessive increases in heart rate with standing and in improving the symptoms of orthostatic intolerance in patients with this disorder.

DETAILED DESCRIPTION:
This trial is designed to study the effects of various mechanistically unique medications in controlling excessive increases in heart rate with standing and in improving the symptoms of orthostatic intolerance in patients with this disorder.

Pilot drug trials are 4h in duration from ~9am -1pm. Different short-acting medications will be used to determine their acute hemodynamic effects in patients with orthostatic intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic symptoms (> 6 months) with standing upright

Exclusion Criteria:

* Obvious cause of hypovolemia or drugs that could worsen tachycardia
* Chronic severe medical conditions such as cancer or ischemic heart disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 1997-04 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Increase in heart rate with standing | 1-4 hours

SECONDARY OUTCOMES:
Sitting heart rate | 1-4 hours
Standing heart rate | 1-4 hours
Blood pressure | 1-4 hours
Decrease in blood pressure with standing | 1-4 hours
Orthostatic symptoms score | Baseline, 2h, 4h

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Autonomic Dysfunction Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Raj SR, Black BK, Biaggioni I, Harris PA, Robertson D. Acetylcholinesterase inhibition improves tachycardia in postural tachycardia syndrome. Circulation. 2005 May 31;111(21):2734-40. doi: 10.1161/CIRCULATIONAHA.104.497594. Epub 2005 May 23. PMID 15911704
- [Result] Raj SR, Black BK, Biaggioni I, Paranjape SY, Ramirez M, Dupont WD, Robertson D. Propranolol decreases tachycardia and improves symptoms in the postural tachycardia syndrome: less is more. Circulation. 2009 Sep 1;120(9):725-34. doi: 10.1161/CIRCULATIONAHA.108.846501. Epub 2009 Aug 17. PMID 19687359
- [Derived] Smith EC, Diedrich A, Raj SR, Gamboa A, Shibao CA, Black BK, Peltier A, Paranjape SY, Biaggioni I, Okamoto LE. Splanchnic Venous Compression Enhances the Effects of ss-Blockade in the Treatment of Postural Tachycardia Syndrome. J Am Heart Assoc. 2020 Jul 21;9(14):e016196. doi: 10.1161/JAHA.120.016196. Epub 2020 Jul 16. PMID 32673517
- [Derived] Nwazue VC, Paranjape SY, Black BK, Biaggioni I, Diedrich A, Dupont WD, Robertson D, Raj SR. Postural tachycardia syndrome and inappropriate sinus tachycardia: role of autonomic modulation and sinus node automaticity. J Am Heart Assoc. 2014 Apr 10;3(2):e000700. doi: 10.1161/JAHA.113.000700. PMID 24721800
- [Derived] Nwazue VC, Arnold AC, Raj V, Black BK, Biaggioni I, Paranjape SY, Orozco C, Dupont WD, Robertson D, Raj SR. Understanding the placebo effect in clinical trials for postural tachycardia syndrome. Clin Exp Pharmacol Physiol. 2014 May;41(5):325-30. doi: 10.1111/1440-1681.12221. PMID 24606242
- [Derived] Green EA, Black BK, Biaggioni I, Paranjape SY, Bagai K, Shibao C, Okoye MC, Dupont WD, Robertson D, Raj SR. Melatonin reduces tachycardia in postural tachycardia syndrome: a randomized, crossover trial. Cardiovasc Ther. 2014 Jun;32(3):105-12. doi: 10.1111/1755-5922.12067. PMID 24495468
- [Derived] Mar PL, Raj V, Black BK, Biaggioni I, Shibao CA, Paranjape SY, Dupont WD, Robertson D, Raj SR. Acute hemodynamic effects of a selective serotonin reuptake inhibitor in postural tachycardia syndrome: a randomized, crossover trial. J Psychopharmacol. 2014 Feb;28(2):155-61. doi: 10.1177/0269881113512911. Epub 2013 Nov 13. PMID 24227635
- [Derived] Green EA, Raj V, Shibao CA, Biaggioni I, Black BK, Dupont WD, Robertson D, Raj SR. Effects of norepinephrine reuptake inhibition on postural tachycardia syndrome. J Am Heart Assoc. 2013 Sep 3;2(5):e000395. doi: 10.1161/JAHA.113.000395. PMID 24002370
- See also: Vanderbilt University Autonomic Dysfunction Center website — https://www.vumc.org/autonomic-dysfunction-center/vanderbilt-autonomic-dysfunction